CLINICAL TRIAL: NCT06246526
Title: Real-World Efficacy of Evoke® Closed-loop Spinal Cord Stimulation (CL-SCS) Therapy in Chronic Pain Patients (ULTRA).
Acronym: ULTRA
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Francis Hospital (Other)
Collaborators: Saluda Medical Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ULTRA Protocol 1.0
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Pain; Chronic Pain; Neuropathic Pain
Keywords: Saluda; Spinal Cord Stimulation
MeSH Terms: conditions — Pain; Chronic Pain; Neuralgia | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Evoke — The Saluda Medical Evoke® CL-SCS System (Evoke System). The Evoke System measures and records spinal cord (SC) activation resulting from stimulation via evoked compound action potentials (ECAPs). The Evoke System can be programmed to provide ECAP-controlled, closed-loop SCS or open-loop, fixed-output (traditional) SCS; ECAPs may be measured and recorded in either stimulation mode.
  Other Names: Spinal Cord Stimulation

SUMMARY:
This observational, prospective data collection is designed to evaluate the efficacy of CL-SCS therapy in real-world patients suffering from chronic pain.

ELIGIBILITY:
Inclusion Criteria:

Be 18 years of age or older at the time of enrollment.

Diagnosed with chronic, intractable pain of the trunk and/or limbs, which has been refractory to conservative therapy for a minimum of 6 months.

Subject has a minimum Visual Analog Scale (VAS) score of 60 mm or higher (where 100 mm indicates the worst imaginable pain) at baseline.

Be an appropriate candidate for the surgical procedures required in this study based on the clinical judgment of the implanting physician.

Be willing and capable of giving informed consent.

Be willing and able to comply with study-related requirements, procedures, and visits.

Exclusion Criteria:

Subject is pregnant or nursing.

Have a medical condition or pain in other area(s), not intended to be treated with SCS, that could interfere with study procedures, as determined by the Investigator.

Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance of intervention, and/or ability to evaluate treatment outcomes.

Have an existing drug pump and/or SCS system or another active implantable device such as a pacemaker, deep brain stimulator (DBS), or sacral nerve stimulator (SNS).

Have prior experience with SCS.

Be concomitantly participating in another clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS - Visual Analog Scale | Baseline to 12 months

SECONDARY OUTCOMES:
PROMIS-29 | Baseline to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Deer, MD, Principal Investigator — Spine and Nerve Center of Saint Francis Hospital
Locations (1):
- The Spine and Nerve Center of Saint Francis Hospital, Charleston, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No